CLINICAL TRIAL: NCT05063552
Title: A Phase II/III Trial of Chemotherapy + Cetuximab vs Chemotherapy + Bevacizumab vs Atezolizumab + Bevacizumab Following Progression on Immune Checkpoint Inhibition in Recurrent/Metastatic Head and Neck Cancers
Brief Title: Testing the Use of Investigational Drugs Atezolizumab and/or Bevacizumab With or Without Standard Chemotherapy in the Second-Line Treatment of Advanced-Stage Head and Neck Cancers
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-10021; NCI-2021-10021 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA3202 (Other: ECOG-ACRIN Cancer Research Group); EA3202 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2021-09-30; First posted 2021-10-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Lip and Oral Cavity Carcinoma; Metastatic Nasal Cavity Squamous Cell Carcinoma; Metastatic Nasopharyngeal Squamous Cell Carcinoma; Metastatic Pharyngeal Squamous Cell Carcinoma; Metastatic Sinonasal Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Nasopharyngeal Squamous Cell Carcinoma; Recurrent Pharyngeal Squamous Cell Carcinoma; Recurrent Sinonasal Squamous Cell Carcinoma; Stage IV Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Nasopharyngeal Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Sinonasal Cancer AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Lymphoid Interstitial Pneumonia; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Carcinoma; Carcinoma | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Carboplatin; Cetuximab; (225)Ac-DOTA-c(RGDyK); Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase II, Arm A (Cetuximab, Docetaxel, Cisplatin, Carboplatin) (Active Comparator): Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 of each cycle, docetaxel IV over 1 hour on day 1 or days 1 and 8 of each cycle, and cisplatin IV or carboplatin IV on day 1 or days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 or days 1 and 15 of each cycle of maintenance therapy. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or MRI throughout the trial. Patients may undergo ECHO during screening. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Biological: Cetuximab; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Phase II, Arm B(Docetaxel, Cisplatin/Carboplatin, Bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 of each cycle, docetaxel IV over 1 hour on day 1 or days 1 and 8 of each cycle, and cisplatin IV or carboplatin IV on day 1 or days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab IV over 30-60 minutes on day 1 of each cycle of maintenance therapy. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or MRI throughout the trial. Patients may undergo ECHO during screening. Patients undergo blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Phase II, Arm C (Bevacizumab, Atezolizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1 and atezolizumab IV over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or MRI throughout the trial. Patients may undergo ECHO during screening. Patients undergo blood sample collection throughout the study.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Phase III, Arm A (Cetuximab, Docetaxel, Cisplatin/Carboplatin) (Experimental): Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 of each cycle, docetaxel IV over 1 hour on day 1 or days 1 and 8 of each cycle, and cisplatin IV or carboplatin IV on day 1 or days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 or days 1 and 15 of each cycle of maintenance therapy. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or MRI throughout the trial. Patients may undergo ECHO during screening. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Biological: Cetuximab; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Phase III, Arm B (Chemotherapy, Bevacizumab, Atezolizumab) (Experimental): Patients receive treatment as in Arm B or C above based on results of the Phase II trial.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Phase II, Arm C (Bevacizumab, Atezolizumab); Phase III, Arm B (Chemotherapy, Bevacizumab, Atezolizumab)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Phase II, Arm B(Docetaxel, Cisplatin/Carboplatin, Bevacizumab); Phase II, Arm C (Bevacizumab, Atezolizumab); Phase III, Arm B (Chemotherapy, Bevacizumab, Atezolizumab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Phase II, Arm A (Cetuximab, Docetaxel, Cisplatin, Carboplatin); Phase II, Arm B(Docetaxel, Cisplatin/Carboplatin, Bevacizumab); Phase II, Arm C (Bevacizumab, Atezolizumab); Phase III, Arm A (Cetuximab, Docetaxel, Cisplatin/Carboplatin)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Phase II, Arm A (Cetuximab, Docetaxel, Cisplatin, Carboplatin); Phase II, Arm B(Docetaxel, Cisplatin/Carboplatin, Bevacizumab); Phase III, Arm A (Cetuximab, Docetaxel, Cisplatin/Carboplatin); Phase III, Arm B (Chemotherapy, Bevacizumab, Atezolizumab)
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Phase II, Arm A (Cetuximab, Docetaxel, Cisplatin, Carboplatin); Phase III, Arm A (Cetuximab, Docetaxel, Cisplatin/Carboplatin)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Phase II, Arm A (Cetuximab, Docetaxel, Cisplatin, Carboplatin); Phase II, Arm B(Docetaxel, Cisplatin/Carboplatin, Bevacizumab); Phase III, Arm A (Cetuximab, Docetaxel, Cisplatin/Carboplatin); Phase III, Arm B (Chemotherapy, Bevacizumab, Atezolizumab)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Phase II, Arm A (Cetuximab, Docetaxel, Cisplatin, Carboplatin); Phase II, Arm B(Docetaxel, Cisplatin/Carboplatin, Bevacizumab); Phase III, Arm A (Cetuximab, Docetaxel, Cisplatin/Carboplatin); Phase III, Arm B (Chemotherapy, Bevacizumab, Atezolizumab)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II/III compares the standard therapy (chemotherapy plus cetuximab) versus adding bevacizumab to standard chemotherapy, versus combination of just bevacizumab and atezolizumab in treating patients with head and neck cancer that has spread to other places in the body (metastatic or advanced stage) or has come back after prior treatment (recurrent). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Cetuximab is in a class of medications called monoclonal antibodies. It binds to a protein called EGFR, which is found on some types of cancer cells. This may help keep cancer cells from growing. Cisplatin and carboplatin are in a class of chemotherapy medications known as platinum-containing compounds. They work by killing, stopping, or slowing the growth of cancer cells. Docetaxel is in a class of chemotherapy medications called taxanes. It stops cancer cells from growing and dividing and may kill them. The addition of bevacizumab to standard chemotherapy or combination therapy with bevacizumab and atezolizumab may be better than standard chemotherapy plus cetuximab in treating patients with recurrent/metastatic head and neck cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) of patients treated with chemotherapy plus cetuximab, chemotherapy plus bevacizumab, and atezolizumab plus bevacizumab. (Phase II) II. To evaluate the overall survival (OS) of patients treated with chemotherapy plus cetuximab to the superior arm from the phase II portion of the protocol. (Phase III)

SECONDARY OBJECTIVES:

I. To evaluate the OS for the subset of patients with high PD-L1 expression, defined as combined positive score (CPS) >= 20% on all arms of treatment.

II. To evaluate the toxicity of each arm of treatment.

IMAGING OBJECTIVES:

I. To establish the correlation between fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET) and computed tomography (CT) neck imaging biomarkers (maximum standard uptake value [SUVmax], metabolic tumor volume [MTV], total lesion glycolysis [TLG], tumor volume) and expression of PD-L1 expression (Low versus high, defined as CPS < 20 versus CPS >= 20).

II. To determine if 18FDG-PET/CT and CT neck imaging biomarkers at baseline will predict treatment response at nine to twelve weeks post the initiation of treatment, PFS, and OS.

EXPLORATORY OBJECTIVE:

I. To establish the correlation between 18F-FDG PET and CT neck radiomics features and PD-L1 expressions (Low versus high - defined as CPS < 20 versus CPS >= 20).

OUTLINE: This is a randomized phase II trial followed by a randomized phase III trial.

PHASE II: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive cetuximab intravenously (IV) over 60-120 minutes on days 1, 8, and 15 of each cycle, docetaxel IV over 1 hour on day 1 or days 1 and 8 of each cycle, and cisplatin IV or carboplatin IV on day 1 or days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 or days 1 and 15 of each cycle of maintenance therapy. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or magnetic resonance imaging (MRI) throughout the trial. Patients may undergo echocardiography (ECHO) during screening.

ARM B: Patients receive bevacizumab IV over 30-90 minutes on day 1 of each cycle, docetaxel IV over 1 hour on day 1 or days 1 and 8 of each cycle, and cisplatin IV or carboplatin IV on day 1 or days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab IV over 30-60 minutes on day 1 of each cycle of maintenance therapy. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or MRI throughout the trial. Patients may undergo ECHO during screening.

ARM C: Patients receive bevacizumab IV over 30-90 minutes on day 1 and atezolizumab IV over 30-60 minutes on day 1 of each cycle. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or MRI throughout the trial. Patients may undergo ECHO during screening.

PHASE III: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 of each cycle, docetaxel IV over 1 hour on day 1 or days 1 and 8 of each cycle, and cisplatin IV or carboplatin IV on day 1 or days 1 and 8 of each cycle. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 or days 1 and 15 of each cycle of maintenance therapy. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo a CT scan, a PET scan, and/or MRI throughout the trial. Patients may undergo ECHO during screening.

ARM B: Patients receive treatment as in Arm B or C above based on results of the Phase II trial.

Patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months if patient is < 2 years from randomization and every 6 months if patient is 2-5 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed squamous cell carcinoma of the head and neck (HNSCC) (excluding squamous cell carcinoma [SCC] of salivary glands, Epstein-Barr virus [EBV]-associated nasopharynx and skin)
* Patient must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Measurements must be obtained within 4 weeks prior to randomization
* Patient must be >= 18 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must have disease progression after prior therapy with an immune checkpoint inhibitor (ICI) in the first-line setting for recurrent/metastatic disease. Patient must have received first-line immune checkpoint inhibition for at least 6 weeks. Patients who have recurred or progressed within 12 weeks of immune checkpoint inhibition administered in the definitive setting for locally advanced disease (for e.g., in the context of a clinical trial) will also be eligible if local therapies are not feasible
* Prior combination immunotherapies are permitted, but patient must not have had prior antiangiogenic treatment (e.g., bevacizumab, ziv-aflibercept, ramucirumab, sorafenib, sunitinib, pazopanib, regorafenib, lenvatinib, etc.). Patient must have completed any prior investigational therapy at least 28 days prior to randomization.

  * NOTE: Patients who received platinum/taxanes in the locally-advanced or recurrent/metastatic setting and did not progress for at least 4 months thereafter, will be eligible for this study. Patients who received cetuximab in the locally-advanced setting and did not progress for at least 4 months thereafter, will also be eligible for this study
* Patient must not have a history of >= grade 3 immune-related adverse event on prior ICI therapy (except those that could be managed with steroids [e.g., dermatologic toxicity, asymptomatic elevation of pancreatic enzymes, etc.]) and ICI could eventually be resumed. Patients who developed grade 3 endocrinopathies but are now stable on hormone supplementation and/or a daily prednisone dose of =< 10 mg (or equivalent doses of another glucocorticoid), will be permitted on this trial
* Patient must not have a history of PD-1 inhibitor-induced hyper-progression, defined as 100% increase in tumor burden within 8 weeks (or 50% within 4 weeks) of initiating ICI and associated with clinical deterioration
* Patient must not have any of the following criteria due to the possibility of increased risk for tumor bleeding with bevacizumab therapy:

  * Prior carotid bleeding,
  * Tumors that invade major vessels (e.g., the carotid) as shown unequivocally by imaging studies,
  * Central (e.g., within 2 cm from the hilum) lung metastases that are cavitary as shown unequivocally by imaging studies,
  * Any prior history of bleeding related to the current head and neck cancer,
  * History of gross hemoptysis (bright red blood of 1/2 teaspoon or more per episode of coughing) within 3 months prior to randomization
* Patient must not have uncontrolled hypertension, a history of hypertensive crisis or hypertensive encephalopathy, or a history of grade 4 thromboembolism
* Patient must not have a history of coagulopathy or hemorrhagic disorders
* Patient must not have a history of thrombosis (e.g., pulmonary embolism or deep venous thrombosis) currently requiring therapeutic anticoagulation (prophylactic use of anticoagulation is allowed)
* Patient must not be receiving chronic daily treatment with aspirin (> 325 mg/day) or non-steroidal anti-inflammatory agents (NSAID's) known to inhibit platelet function. The use of anti-platelet agents [e.g., dipyridamole (Persatine), ticlopidine (Ticlid), clopidogrel (Plavix)] is allowed only if patient is not receiving concurrent aspirin or NSAID's known to inhibit platelet function
* Patient must have PD-L1 expression >= 1% by CPS in the tumor and/or immune cells

  * NOTE: Enrolling centers should test for PD-L1 CPS preferably using the SP263 assay. Where this is not feasible, using their preferred Clinical Laboratory Improvement Act (CLIA)-certified or similar assay will be accepted. It is preferred for standard of care (SOC) PD-L1 assessments to be done on post-first line ICI samples if available, but SOC PD-L1 assessments on pre-ICI samples will be accepted for eligibility
* Patient must not have a severe infection within 4 weeks prior to randomization, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. Patients must not have active tuberculosis
* Patient must not have a history of non-infectious pneumonitis requiring steroids at doses greater than or equal to 10 mg per day of prednisone or the equivalent on first line immunotherapy
* Patient must not have a history of solid organ transplantation or stem-cell transplant
* Patient must not be on immunosuppressive medication within 7 days prior to randomization except for: intranasal, inhaled, or topical steroids, local steroid injection, systemic corticosteroids at doses less than or equal to 10 mg per day of prednisone or the equivalent, or steroids used as premedication for hypersensitivity reactions
* Patient must not have an active autoimmune disease that requires systemic treatment within 2 years prior to randomization. Patients who are receiving replacement therapy for adrenal or pituitary insufficiency will not be excluded
* Patient must not have had a severe hypersensitivity reaction to any of the drug components used on this protocol or to chimeric or humanized antibodies or fusion proteins
* Patient must not have received any live vaccine within 30 days prior to randomization and while participating in the study (and continue for 5 months after the last dose of atezolizumab on Arm C). Live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine. Patients are permitted to receive inactivated vaccines and any non-live vaccines including those for the seasonal influenza and coronavirus disease 2019 (COVID-19) (Note: intranasal influenza vaccines, such as Flu-Mist [registered trademark] are live attenuated vaccines and are not allowed). If possible, it is recommended to separate study drug administration from vaccine administration by about a week (primarily, in order to minimize an overlap of adverse events
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patients must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 2 months after the last dose of treatment for patients assigned to Arm A and for 6 months after the last dose of protocol treatment for patients assigned to Arms B or C.

  * NOTE: Patients must also not breastfeed while on treatment and for 2 months after the last dose of treatment for patients assigned to Arm A and for 6 months after the last dose of treatment for patients assigned to Arms B or C
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Leukocytes >= 3,000/mcL (must be obtained =< 14 days prior to protocol randomization)
* Absolute neutrophil count (ANC) >= 1,500/mcL (must be obtained =< 14 days prior to protocol randomization)
* Platelets >= 100,000/mcL (must be obtained =< 14 days prior to protocol randomization)
* Hemoglobin (Hgb) > 9 g/dL (must be obtained =< 14 days prior to protocol randomization) (Note: Patient may be transfused to meet this criteria)
* Total bilirubin =< 2.0 x institutional upper limit of normal (ULN) (=< 5.0 x institutional ULN if hepatic metastases present or =< 3 x ULN for patients with known Gilbert's disease) (must be obtained =< 14 days prior to protocol randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (< 5.0 x institutional ULN if hepatic metastases present) (must be obtained =< 14 days prior to protocol randomization)
* Alkaline phosphatase < 2.5 x institutional ULN (< 5.0 x institutional ULN if hepatic or bone metastases present) (must be obtained =< 14 days prior to protocol randomization)
* Creatinine =< 1.5 x institutional ULN (must be obtained =< 14 days prior to protocol randomization)
* Patients with uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN) must have their calcium levels corrected prior to randomization
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. Patients must not have untreated brain metastases or leptomeningeal disease
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients must not have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients may have indwelling catheters (e.g., PleurX [registered trademark])
* Patient must not have significant cardiovascular disease (such as New York Heart Association class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to randomization, or unstable arrhythmia or unstable angina at the time of randomization
* Patient must not receive any other chemotherapy, immunotherapy, antitumor hormonal therapy (excluding contraceptives and replacement steroids), radiation therapy, or experimental medications while on protocol treatment. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to randomization and patients must be recovered from the effects of radiation (there is no required minimum recovery period
* Patient must not have had a surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to randomization, or anticipation of need for major surgical procedure while on protocol treatment
* Patient must not have any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of the agents used in this protocol, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Patient must not have a history of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess, or active GI bleeding within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Phase II) | Time from treatment initiation until disease progression or death, assessed up to 5 years from randomization
Overall survival (OS) (Phase III) | Time from treatment initiation until death from any cause, assessed up to 5 years from randomization
  Will be compared using a stratified log rank test.

SECONDARY OUTCOMES:
OS in the subset of patients with high PD-L1 expression (Phase III) | Up to 5 years from randomization
  The interaction of PD-L1 by treatment will also be evaluated in a Cox proportional hazards model.
Incidence of adverse events (Phase III) | Up to 30 days after completion of treatment
Correlation between fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET) and computed tomography (CT) neck imaging biomarkers | Up to 5 years from randomization
  The two-sample t-test will be used to compare the difference of baseline 18F -FDG PET /CT imaging biomarkers (maximum standardized uptake value [SUVmax], metabolic tumor volume [MTV], total lesion glycolysis [TLG], tumor volume) between low and high expression of PD-L1.
Prediction of treatment response | Baseline up to 12 weeks
  Determined by 18FDG-PET/CT and CT neck imaging biomarkers. To determine if 18FDG-PET/CT and CT neck imaging biomarkers at baseline will predict treatment response at nine to twelve weeks post-treatment, PFS, and OS Logistic regression model will be fit to assess the association of the 18F -FDG PET /CT imaging biomarkers (e.g., SUVmax, MTV, TLG, tumor heterogeneity, tumor volume) with binary treatment response at 9-12 weeks post treatment. Cox proportional hazards models will be fit to assess the association of 18F -FDG PET /CT imaging biomarkers with time-to-event outcomes (PFS or OS).

OTHER OUTCOMES:
Correlation between 18F-FDG PET and CT neck radiomics features and expression of PD-L1 expression | Up to 5 years from randomization
  The imaging textural features from radiomics analysis will be associated with the dichotomized PD-L1 expressions. First, proper transformation will be applied to the textural features as needed to address the distribution skewness. Second, Pearson or Spearman rank correlations will be calculated between all pairs of textural features to identify highly correlated features. Third, to address overfitting and high collinearity, machine learning techniques (e.g., LASSO or XGBoost) will be employed for feature selection during the association analysis with PD-L1 expressions.

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Bhatia, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (172):
- United States (172):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Contra Costa Regional Medical Center, Martinez, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Mercy Hospital, Coon Rapids, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center in Greenville/UPMC Horizon, Greenville, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Covenant Health Cancer Centers, Knoxville, Tennessee
  - Covenant Health Cancer Centers - West, Knoxville, Tennessee
  - Covenant Health Oncology Group - Lenoir City, Lenoir City, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Covenant Health Oncology Group - Oak Ridge, Oak Ridge, Tennessee
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-03-13): https://cdn.clinicaltrials.gov/large-docs/52/NCT05063552/ICF_000.pdf